CLINICAL TRIAL: NCT01043536
Title: Dose Escalation Radiotherapy With Modulation of Intensity and Integrated Boost in Association With a Temozolomide in the Treatment of Glioblastoma
Brief Title: Dose Escalation Radiotherapy With Modulation of Intensity and Integrated Boost (SIB-IMRT) in the Treatment of Glioblastomas in Adults
Acronym: SIB-IMRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0244-1blni08 / 009.020
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Glioblastoma
Keywords: IMRT; Radiotherapy escalation dose; glioblastoma; escalation radiotherapy dose
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiotherapy + temozolomide (Experimental): Radiotherapy:
  dose given at PTV-g will be 70 Gy/28 fractions level 1 75 Gy/30 fractions level 2 80 Gy/32 fractions level 3
  dose given at PTV-a will be 56 Gy/28 fractions level 1 60 Gy/30 fractions level 2 60.8 Gy/32 fractions level 3
  Chemotherapy:
  temozolomide given at the dose of 75mg/m2
  Interventions: Radiation: radiotherapy; Drug: temozolomide

INTERVENTIONS:
Radiation: radiotherapy — patients will receive from 6 to 7 weeks 5 days a week radiations. The dose of radiation will depend on the level they will be included.
Drug: temozolomide — patient will receive whatever the level 7 days a week, temozolomide at the dose of 75mg/m2 during radiotherapy period. They will then follow one month after the end the radiochemotherapy an adjuvant treatment corresponding to a 5 days treatments of temozolomide at the dose of 200mg/m2 every 28 days.

SUMMARY:
The main goal of this study is to evaluate and to determine the dose of a highly accurate irradiation (allowing to increase the dose delivered while restricting the risk of complication) in association with temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of glioblastoma (WHO grade IV astrocytoma)
* Diagnosis must be obtained by a stereotactic or surgical biopsy
* Age between 18 and 70
* Total or partial surgical resection deemed as not possible by a neurosurgeon
* OMS performance status 0 or 1
* Adequate blood function : absolute neutrophil count > 1.5 x 109/L, platelets count > 100 x 109/L platelets;
* Adequate liver function: bilirubin < 1.5 ULN (upper limit of normal), ALT and AST < 3 ULN,
* Adequate renal function: creatinine < 1.5 ULN
* Patient must have been informed and must have signed the specific informed consent form.

Exclusion Criteria:

* other malignancy histology
* resection of the brain tumor complete on MRI exploration
* patient unable to give informed consent
* patient presenting counter-indication to MRI exploration
* patient must not have received neither radiotherapy nor chemotherapy for that affection
* concomitant malignancy
* patient already enrolled in another biomedical study with an experimental molecule
* pregnant, nursing woman, or without contraception
* private individuals of freedom or under tutelage (including legal guardianship)
* psychiatric, behavioural disorders or geographical situation precluding the administration or follow-up of the protocol (including claustrophobia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine the OTR (optimal tolerated regimen) of radiotherapy administered in combination with temozolomide as first-line therapy in patients with de novo glioblastoma | 3 months after the start of the radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Truc, MD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- Centre Georges François Leclerc, Dijon, Bourgogne-Franche-Comté, France